CLINICAL TRIAL: NCT02534961
Title: Prophylactic Administration of Antibiotics Before Radiofrequency Ablation for Hepatocellular Carcinoma: A Randomized Trial
Brief Title: Prophylactic Antibiotics Before RFA for HCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-01-003B
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Radiofrequency ablation; Antibiotics
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prophylactic antibiotics group (Active Comparator): Patients in the prophylactic group will receive antibiotic treatment right after randomization with intravenous cefazolin 2 g (3 g for patients weighing ≥120 kg) within 60 minutes before ablation therapy.
  Interventions: Drug: Cefazolin
- on-demand antibiotics group (No Intervention): Patients in the on-demand group will receive antibiotic therapy only when infection will be suspected or established.

INTERVENTIONS:
Drug: Cefazolin — Patients in the prophylactic group will receive antibiotic treatment right after randomization with intravenous cefazolin 2 g (3 g for patients weighing ≥120 kg) within 60 minutes before ablation therapy. Patients in the on-demand group will receive antibiotic therapy only when infection will be suspected or established. Antibiotics will be changed according to the antibiotic sensitivity test of cultured microorganisms.
  Arms: prophylactic antibiotics group

SUMMARY:
This randomized prospective study aims to investigate whether prophylactic administration of antibiotics has an influence on inflammatory markers, liver function test results, or the incidence of post-procedural infection in patients with hepatocellular carcinoma (HCC) undergoing radiofrequency ablation (RFA).

DETAILED DESCRIPTION:
Patients

1. This cohort study will prospectively enroll HCC patients undergoing RFA in Taipei Veterans General Hospital and Taipei Medical University Hospital.
2. The diagnosis of HCC is established by histology or on the basis of the findings of typical radiologic features in a 4-phase multidetector computed tomography (CT)scan or dynamic contrast-enhanced magnetic resonance imaging (MRI).
3. Inclusion criteria: tumor size less than 5 cm without extra-hepatic metastasis; the number of tumor was 3 or less; Child Pugh classification of liver function are grade A or B; and the absence of other major diseases that might complicate RFA.
4. Patients will be excluded from the study if they meet the following criteria. First, the patient's age is younger than 20 years or older than 80 years. Second, the patients have a terminal illness of any major organ system, like heart failure, uremia, chronic obstructive pulmonary disease, or non-hepatic malignancy. Third, the patients have received antibiotics within the last 2 weeks. Patients will be subsequently excluded when initial bacteriological sampling turned out positive (occult infection).
5. After disinfection of the skin surface and induction of local anesthesia with 1% lidocaine, RFA will be performed with real-time ultrasonography guidance, and the RF electrode will be advanced into the tumor. RFA device will be used the Cool-Tip Radiofrequency System (Radionics, Burlington, MA). With the Cool-Tip device, treatment will be performed with a single (2- or 3-cm active tip) needle electrode. Each tumor has 1-4 ablations per session, depending on the tumor size. If the tumor is adjacent to hollow viscera and can not be displaced with a safe margin of at least 2 cm by positioning the patient in an oblique or lateral position, 5% dextrose will be intraperitoneally instilled around the liver to displace the hollow viscera.
6. After RFA, all patients will undergo immediate follow-up ultrasonography to evaluate the possibility of bleeding or fluid accumulation. Dynamic CT scan or MRI will be done one month after all of the tumors ablated by RFA. When these will be confirmed residual tumors by showing contrast enhancement during the arterial phase and wash out in venous phase, a second session of RFA will be conducted. If viable tumors persist after two sessions of RFA therapy, treatment will be considered a failure. If no viable tumor is detected, the patient will be regularly followed-up with abdominal sonography every 3 months.
7. Tumor recurrence is suspected if there is elevated serum AFP level or new lesion detected by surveillance ultrasonography. These would be confirmed by dynamic CT or MRI. Local recurrence is defined as tumor recurrence at the same segment of a previous tumor site, while intra-hepatic distant recurrence is diagnosed when a new lesion occurs in a different segment of a previously treated tumor.

Randomization Patients who fulfilled the inclusion criteria will be immediately randomized to the two treatment groups by using consecutively numbered envelopes that contained the treatment assignments, which were generated by a computer-allocated random digit number, in a 1:1 ratio. Patients in the prophylactic group will receive antibiotic treatment right after randomization with intravenous cefazolin 2 g (3 g for patients weighing ≥120 kg) within 60 minutes before ablation therapy. Patients in the on-demand group will receive antibiotic therapy only when infection will be suspected or established. Antibiotics will be changed according to the antibiotic sensitivity test of cultured microorganisms.

Infection Assessment All patients will be closely monitored with special emphasis on the detection of bacterial infection through the hospitalization period. A careful physical examination, complete white blood cell count, chest radiography, urine sediment, urine culture, ascitic fluid neutrophil count and culture (if available), and blood culture will be routinely performed before randomization. Physical examination will be performed at least once per day during hospitalization. If a new infection is suspected, the same procedures to assess infection would be performed at admission. New infections are suspected when there is fever (>38°C), hypothermia (<36°C), unexpected hemodynamic instability, tachypnea, new onset of chest symptoms, dysuria, abdominal pain, distention, as well as alteration of mental state. A central venous catheter or urinary catheter would be inserted only when clinically indicated.

Clinical Assessment and Follow-up Body temperature will be measured every 6 hour for 72 hour. Acetaminophen at 500 mg will be used when patients complain of pain or have a high grade fever over 39°C after the procedure. The numbers of peripheral blood leukocytes, as well as levels of serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), creatinine, C-reactive protein (CRP) and infection signs as above descriptions will be determined before, and at 24 hour, 3-7 day and 4 week after ablation therapy. Dynamic CT scan or MRI will be done one month after all of the tumors ablated by RFA in order to estimate the effectiveness of RFA or HCC, and whether liver abscess, cholangitis, cholangitis and peritonitis will be present. If a new infection is suspected within one month after RFA, Dynamic CT scan or MRI will be done immediately. Post-procedure infection is defined on the Guideline for Prevention of Surgical Site Infection, 1999, Centers for Disease Control and Prevention (CDC).

Safety Assessment and Adverse Events Adverse events will be recorded by the investigators during hospitalization or at the 4-week out-patient follow-up visit.

Statistical Analysis Pearson chi-square analysis or Fisher's exact test will be used to compare categorical variables, while the Mann-Whitney U-test would be used to compare continuous variables.

Variables with statistical significance (p<0.05) or proximate to it (p<0.1) by univariate analysis underwent multivariate analysis using a Cox's forward stepwise logistic regression model. A two-tailed p value <0.05 is considered statistically significant. All statistical analyses will be performed using the Statistical Package for Social Sciences (SPSS 19.0 for Windows, SPSS. Inc., Chicago, IL, USA).

The infection rate of patients with HCC after RFA, without special emphasis on antibiotics treatment, is 1.5-3%. Estimates of sample size are based on a infection rate assumed to be 1% for the prophylactic antibiotics group and 5% for the on-demand antibiotics group. The type I (alpha) error and type II (beta) error are set to 0.05 and 0.2, respectively. The sample size needed is estimated to be at least 282 patients per group. Taking into account an expected dropout or missing data rate of 5%, the sample size needed is estimated to be at least 594 patients. Consequently, we plan to enroll a total of 600 patients in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCC and underwent RFA
2. With tumor size less than 5 cm without extra-hepatic metastasis;

2. The number of tumor was 3 or less; 3. Child Pugh classification of liver function are grade A or B; 4. Absence of other major diseases that might complicate RFA.

Exclusion Criteria:

1. Age is younger than 20 years or older than 80 years.
2. Patients have a terminal illness of any major organ system, like heart failure, uremia, chronic obstructive pulmonary disease, or non-hepatic malignancy.
3. Patients have received antibiotics within the last 2 weeks. Patients will be subsequently excluded when initial bacteriological sampling turned out positive (occult infection).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Infection after radiofrequency ablation | within 4 weeks after radiofrequency ablation
  Body temperature will be measured every 6 hour for 72 hour. Acetaminophen at 500 mg will be used when patients complain of pain or have a high grade fever over 39°C after the procedure. The numbers of peripheral blood leukocytes, as well as levels of serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), creatinine, C-reactive protein (CRP) and infection signs as above descriptions will be determined before, and at 24 hour, 3-7 day and 4 week after ablation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Wei Su, MD & PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Division of Gastroenterology, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan